CLINICAL TRIAL: NCT01661673
Title: Safety, Tolerability, Pharmacokinetics, and Effects of EVP-0962 on Cerebral Spinal Fluid Amyloid Concentrations in Healthy Subjects and in Subjects With Mild Cognitive Impairment or Early Alzheimer's Disease
Brief Title: Safety, Tolerability, Pharmacokinetics of EVP-0962 and Effects of EVP-0962 on Cerebral Spinal Fluid Amyloid Concentrations in Healthy Subjects and in Subjects With Mild Cognitive Impairment or Early Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FORUM Pharmaceuticals Inc (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVP-0962-002
Record Dates: First submitted 2012-08-03; First posted 2012-08-09 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Experimental): 10 mg EVP-0962 Orally administered once daily for 14 days
  Interventions: Drug: EVP-0962
- Arm 2 (Experimental): 50 mg EVP-0962 Orally administered once daily for 14 days
  Interventions: Drug: EVP-0962
- Arm 3 (Experimental): 100 mg EVP-0962 Orally administered once daily for 14 days
  Interventions: Drug: EVP-0962
- Arm 4 (Experimental): 200 mg EVP-0962 Orally administered once daily for 14 days
  Interventions: Drug: EVP-0962
- Arm 5 (Placebo Comparator): Placebo orally administered for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EVP-0962 — Arms: 1,2,3,4
  Arms: Arm 1; Arm 2; Arm 3; Arm 4
Drug: Placebo — Arm 5
  Arms: Arm 5

SUMMARY:
This study is being conducted to determine the safety, tolerability, pharmacokinetics, and effects of EVP-0962 on cerebral spinal fluid Amyloid concentrations in healthy subjects and in subjects with mild cognitive impairment or early Alzheimer's disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind, sequential escalating repeat daily dose study conducted in two parts. The first part is being conducted in healthy subjects and will evaluate safety, tolerability, and pharmacokinetics and pharmacodynamics of escalating EVP-0962 doses (10, 50 100 and 200 mg) or matching placebo following once-daily administration for 14 days. The second part will evaluate the safety, tolerability and pharmacokinetics and pharmacodynamics of EVP-0962 following once-daily administration for 14 days in patients with mild cognitive impairment or early Alzheimer's disease at the dose level selected based on the available safety, pharmacokinetics and pharmacodynamics observations in the first part.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Male and female subjects between the ages of 45 to 65 (inclusive) in good health with a BMI of 18-32 kg/m2 and negative urine drug screen of abuse test.
* Part 2: Male and female subjects between the ages of 45 to 85 (inclusive), MRI/CT scans compatible with diagnosis of MCI or early AD, meets the classification of MCI due to AD as defined by the National Institute on Aging-Alzheimer's Association, and a BMI of 18-32 kg/m2(inclusive). Subjects must meet the following Cognitive criteria: Subject Memory Complaint, cognitive impairment in one or more areas, CDR-SB score less than or equal 1.0, MMSE greater than 24, and no impairment in social or occupational functioning.

Exclusion Criteria:

* History of seizure disorder, symptomatic orthostatic hypotension, QTc values greater than 450 ms, positive drug screening tests
* Pregnancy, nursing, (or if fertile female) not willing to utilize birth control measures during study
* C-SSRS suicidal ideation score of 4 or 5
* Unwilling to abstain from vigorous exercise
* Concurrent disease other than MCI or early AD that is attributing to patient's cognitive impairment.
* Lumbar spine X-rays show anatomic contraindications to lumbar puncture
* History of spinal surgery or chronic low back pain
* History of migraine headaches

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-11; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The number of adverse experiences reported by subjects and/or observed by investigator and repeated clinical evaluations of physical examinations, vital signs, 12-lead ECG (electrocardiogram), and lab tests (hematology, chemistry, urinalysis) | Screening (Day-45 to Day -1) through Day 23 (end of study visit)
To measure the rate of synthesis of Amyloid Beta in cerebral spinal fluid of healthy subjects | 0-36 hours post dose
To measure the concentration of Amyloid Beta in cerebral spinal fluid | 0-36 hours post dose

SECONDARY OUTCOMES:
To measure the rate of synthesis of Amyloid Beta and steady-state levels in the cerebral spinal fluid in MCI or early Alzheimer's disease patients | 0-36 hours post dose
To determine single-and repeat-dose EVP-0962 pharmacokinetics in cerebral spinal fluid and plasma | 0-36 hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Glendale Adventist Medical Center, Glendale, California, United States